CLINICAL TRIAL: NCT03915990
Title: Middle Cerebral and Umbilical Arteries Doppler Indices in Pregestational Diabetic Versus Normal Pregnancies and Their Values in Predicting Adverse Neonatal Outcome
Brief Title: Middle Cerebral and Umbilical Arteries Doppler Indices in the Prediction of Adverse Neonatal Outcome Among Diabetic Pregnant Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Moutaz Sherbini, assistant professor (MD) Obs & Gyn., Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 35343332
Record Dates: First submitted 2019-04-12; First posted 2019-04-16 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: diabetes; umbilical artery; middle cerebral artery
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (Other): 60 healthy pregnant women will be included
  Interventions: Diagnostic Test: umbilical and middle cerebral artery Doppler
- controlled diabetics (Active Comparator): 30 diabetic pregnant women with controlled Diabetes (i.e. HbA1C less than 6.5 %)
  Interventions: Diagnostic Test: umbilical and middle cerebral artery Doppler
- uncontrolled diabetics (Active Comparator): 30 diabetic pregnant women with uncontrolled Diabetes (i.e. HbA1C equal or more to 6.5 %)
  Interventions: Diagnostic Test: umbilical and middle cerebral artery Doppler

INTERVENTIONS:
Diagnostic Test: umbilical and middle cerebral artery Doppler — Umbilical and middle cerebral arteries Doppler indices (resistance index and pulsatility index) and Cerebroplacental Doppler ratio will be measured for every patient.

SUMMARY:
120 patients will be included and divided into two groups; Control group that will include 60 healthy pregnant women and Study group that will include 60 pregestational diabetic pregnant patients which furtherly will be subdivided into two groups according to HbA1C levels namely; controlled diabetics ( will include 30 diabetic pregnant women with controlled DM - HbA1C < 6.5 %) and uncontrolled diabetics (will include 30 diabetic pregnant women with uncontrolled DM - HbA1C ≥ 6.5 %). Umbilical and middle cerebral arteries Doppler indices (resistance index and pulsatility index) and Cerebroplacental Doppler ratio will be measured for every patient. The recorded neonatal outcomes will include neonatal birth weight, neonatal blood sugar, Apgar score at 1 & 5 min and neonatal intensive care unit admission.

DETAILED DESCRIPTION:
120 pregnant women (aged from 18- to 40 years old) with singleton healthy living fetus between 34 -37 weeks gestation will be included in the current study and they will be divided into two groups; Control group that will include 60 healthy pregnant women and Study group that will include 60 pregestational diabetic pregnant patients. The latter group will be furtherly subdivided into two groups according to HbA1C levels namely; controlled diabetics (will include 30 diabetic pregnant women with controlled DM - HbA1C < 6.5 %) and uncontrolled diabetics (will include 30 diabetic pregnant women with uncontrolled DM - HbA1C ≥ 6.5 %). The patient will be recruited from the obstetric out-patient clinic and in-patient department (Department of Obstetrics & Gynecology - Kasr El-Aini Hospital - Faculty of Medicine - Cairo University). Diabetic women with either complicated diabetes or any other chronic diseases (e.g., hypertension or renal) will be excluded. Patients with anomalous or IUGR (EFW below the 10th percentile for gestational age) fetuses will be excluded. Patients experienced any pregnancy induced medical disorders, rupture of membranes or oligohydramnios (AFI < the fifth percentile) in the current pregnancy will be also excluded.

Informed consent will be obtained from all participants (to share in the study after describing the aim of the study and the potential hazards) then all participants will be subjected to the following: full history taking, complete Physical Examination (general & local), laboratory investigations (Complete blood picture, liver & kidney functions, Fasting and post prandial blood sugar and HbA1C estimation) and routine obstetric ultrasound (to confirm gestational age, assess fetal weight (EFW) and amniotic fluid index (AFI) and to exclude fetal anomalies. Doppler ultrasonography assessment will be done using the apparatus (SonoAce R3 with Doppler unit and convex linear transducer 3.5 MHZ). As regard umbilical artery (UA) Doppler, all patients will be placed in a semi recumbent position with a left lateral tilt, and then the uterine content will be scanned to select an area of amniotic cavity with several loops of cord. Then using a pulsed wave Doppler on a free loop of cord, the characteristic sound and shape of the umbilical artery will be identified. When the screen showed at least 3 consecutive wave forms of similar height, the image will be frozen and umbilical artery Doppler parameters (Resistance index and pulsatility index) will be estimated. A minimum of 3 separate readings will be averaged before the final values are obtained. Umbilical artery Doppler studies will be avoided during fetal activity and fetal breathing because of effect of fetal breathing movements on waveform variability and recording will be performed during fetal apnea. Abnormal UA Doppler velocimetry will be defined if indices more than 95th centile for gestational age or if diastolic flow is either absent or reversed. As regard middle cerebral artery Doppler (MCA), a transverse view of the fetal brain will be obtained at the level of the biparietal diameter. The transducer will then moved towards the base of the skull at the level of the lesser wing of the sphenoid bone. Using color flow imaging, the middle cerebral artery will be seen as a major lateral branch of the circle of Willis, running anterolaterally at the borderline between the anterior and the middle cerebral fossae. The pulsed Doppler sample gate will then placed on the middle portion of this vessel to obtain flow velocity waveforms. When the screen showed at least 3 consecutive wave forms of similar height, the image will be frozen and middle cerebral artery Doppler parameters (Resistance index & pulsatility index) will be estimated. A minimum of 3 separate readings will be averaged before the final values are obtained. Care should be taken to apply minimal pressure to the maternal abdomen with the transducer, as fetal head compression is associated with alterations of intracranial arterial waveforms. Abnormal MCA Doppler velocimetry will be defined if indices less than 5th centile for gestational age. After fetal birth, the following data will be recorded; neonatal birth weight, neonatal blood sugar, Apgar score at 1and 5 min, the need for transfer to neonatal intensive care unit (NICU). Abnormal perinatal outcomes will included one-min and five-min Apgar scores less than 7, hypoglycemia [blood sugar (BS) less than 50 mg/dL], neonatal intensive care unit (NICU) hospitalization. Women with at least one poor outcome will be categorized in the abnormal neonatal outcome group.

ELIGIBILITY:
Inclusion Criteria:

* Single living pregnancy.
* Gestational age: 34-37 weeks (confirmed by a reliable date for the last menstrual period and 1st trimester ultrasound scan).
* Healthy pregnant women in group 1 (control group).
* History of pregestational DM in group 2 (study group) i.e., patients known to be diabetic before pregnancy whether on diet, oral hypoglycemic drugs or insulin therapy.

Exclusion Criteria:

* Fetal anomalies.
* Any maternal chronic diseases esp. renal disease, epilepsy or CNS lesion.
* Pregnancy induced medical disorders.
* IUGR (EFW below the 10th percentile for gestational age).
* Rupture of membranes or oligohydramnios (AFI < the fifth percentile).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
the diagnostic value of Umbilical artery Doppler indices [Resistance index (RI)& pulsatility index (PI)] in predicting the adverse neonatal outcome among diabetic patients. | 34 -37 weeks gestation (for DOPPLER) and at birth (for neonatal outcomes)
  the sensitivity & the specificity of UA RI & PI in predicting the adverse neonatal outcome among diabetic patients.

SECONDARY OUTCOMES:
he diagnostic value of MCA Doppler indices [Resistance index (RI)& pulsatility index (PI)] in predicting the adverse neonatal outcome among diabetic patients. | 34 -37 weeks gestation (for DOPPLER) and at birth (for neonatal outcomes)
  the sensitivity & the specificity of MCA RI & PI in predicting the adverse neonatal outcome among diabetic patients.

CONTACTS AND LOCATIONS:
Locations (1):
- kasr elainy hospital (Faculty of Medicine - Cairo University), Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No